CLINICAL TRIAL: NCT02181543
Title: Use of Intraoperative Clonidine for Prevention of Postoperative Agitation in Pedriatic Anesthesia With Sevoflurane.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Professor Fernando Figueira Integral Medicine Institute (Other)
Responsible Party: Principal Investigator, Alex Sandro Rolland de Souza, Professor, Professor Fernando Figueira Integral Medicine Institute
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: U1111-1157-8852
Record Dates: First submitted 2014-07-02; First posted 2014-07-04 (Estimated); Last update posted 2017-10-04 (Actual); Status verified 2017-10

CONDITIONS: Is an Only Child
Keywords: Clonidine; Psychomotor agitation; Anesthesia recovery period; Tonsillectomy; Child, preschool
MeSH Terms: conditions — Psychomotor Agitation | interventions — Clonidine

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Clonidine (Experimental): Clonidine 1μg/Kg, IV, single dose, anesthesia intraoperative.
  Interventions: Drug: Clonidine
- No Clonidine (No Intervention): Usual care of Instituto de Medicina Integral Prof. Fernando Figueira.

INTERVENTIONS:
Drug: Clonidine — 1μg/Kg, IV (in the vein) intraoperative. Number of Cycles: single dose.
  Arms: Clonidine

SUMMARY:
The purpose of this study is to determine efficacy of intraoperative clonidine to prevent postoperative agitation in pediatric anesthesia with sevoflurane.

ELIGIBILITY:
Inclusion Criteria:

* Aged 2 - 12 Years.
* Need for tonsillectomy / adenotonsillectomy.
* Physical status of the American Society of Anesthesiologists (ASA) 1, 2 or 3.
* Anestesia geral com sevoflurano.
* Use of Intraoperative dipyrone, 30-50mg/Kg, IV.

Exclusion Criteria:

* Changes in consciousness.
* Neurological Deficit.
* Use of another drug as medication before anesthesia.

Ages: 2 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Actual)
Dates: Start 2013-08 (Actual); Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Postoperative agitation | 6 hours
  Postoperative agitation will be assessed by the Pediatric Anesthesia Emergence Delirium Scale (PAED).

SECONDARY OUTCOMES:
Duration of postoperative agitation | 6 hours
  Time in minutes.
Need for post-anesthetic drugs for treatment of agitation | 6 hours
  Use of any drugs, such as sedatives, opioids, anti-inflammatory or anti-emetic for improvement agitation.
Any occurrence of post-anesthesia accidents: falls, bruises or disconnection of catheters | 6 hours
  If any accident occurs in the recovery room, and postoperative (falls, bruises) disconnection of intravenous catheter or injuries.
Drowsiness | 6 hours
  Clinical evaluation: patient awake, awake, alert or patient under hypnosis.
Parental satisfaction. | 24 hours
  As parents answer the question if you are satisfied with the procedure performed, excluding other problems occurred in the hospital.

CONTACTS AND LOCATIONS:
Overall Officials: Alex SR Souza, PhD, Principal Investigator — Instituto de Medicina Integral Prof. Fernando Figueira (IMIP); Fernando A Souza Júnior, MD, Study Chair — Instituto de Medicina Integral Prof. Fernando Figueira (IMIP); Tania CM Couceiro, MD, Study Chair — Instituto de Medicina Integral Prof. Fernando Figueira (IMIP); Ítalo GM Santos, Student, Study Chair — Instituto de Medicina Integral Prof. Fernando Figueira (IMIP); Luciana C Lima, PhD, Study Director — Instituto de Medicina Integral Prof. Fernando Figueira (IMIP)
Locations (1):
- Instituto de Medicina Integral Prof. Fernando Figueira (IMIP), Recife, Pernambuco, Brazil

REFERENCES:
- [Background] Hudek K. Emergence delirium: a nursing perspective. AORN J. 2009 Mar;89(3):509-16; quiz 517-9. doi: 10.1016/j.aorn.2008.12.026. PMID 19326585
- [Background] Silva LM, Braz LG, Modolo NS. Emergence agitation in pediatric anesthesia: current features. J Pediatr (Rio J). 2008 Mar-Apr;84(2):107-13. doi: 10.2223/JPED.1763. PMID 18372935
- [Result] Kulka PJ, Bressem M, Tryba M. Clonidine prevents sevoflurane-induced agitation in children. Anesth Analg. 2001 Aug;93(2):335-8, 2nd contents page. PMID 11473855
- [Result] Malviya S, Voepel-Lewis T, Ramamurthi RJ, Burke C, Tait AR. Clonidine for the prevention of emergence agitation in young children: efficacy and recovery profile. Paediatr Anaesth. 2006 May;16(5):554-9. doi: 10.1111/j.1460-9592.2006.01818.x. PMID 16677266
- [Result] Fazi L, Jantzen EC, Rose JB, Kurth CD, Watcha MF. A comparison of oral clonidine and oral midazolam as preanesthetic medications in the pediatric tonsillectomy patient. Anesth Analg. 2001 Jan;92(1):56-61. doi: 10.1097/00000539-200101000-00011. PMID 11133600
- [Result] Tazeroualti N, De Groote F, De Hert S, De Ville A, Dierick A, Van der Linden P. Oral clonidine vs midazolam in the prevention of sevoflurane-induced agitation in children. a prospective, randomized, controlled trial. Br J Anaesth. 2007 May;98(5):667-71. doi: 10.1093/bja/aem071. Epub 2007 Apr 7. PMID 17416907
- [Derived] Sousa-Junior FA, Souza ASR, Lima LC, Santos IGM, Menezes LAP, Ratis PAPL, Couceiro TCM. Intraoperative clonidine to prevent postoperative emergence delirium following sevoflurane anesthesia in pediatric patients: a randomized clinical trial. Braz J Anesthesiol. 2021 Jan-Feb;71(1):5-10. doi: 10.1016/j.bjane.2020.12.003. Epub 2020 Dec 25. PMID 33712253
- See also: Instituto de Medicina Integral Prof. Fernando Figueira (IMIP) — http://www.imip.org.br